CLINICAL TRIAL: NCT06138756
Title: A Prospective, Single Arm, Open Label Post Market Study Assessing the Safety and Efficacy of Nerivio for the Treatment of Migraine in Children Under the Age of 12
Brief Title: Acute Treatment of Migraine in Pre-Adolescents: Real-World Analysis of Remote Electrical Neuromodulation (REN)
Status: Completed | Type: Observational
Sponsor: Theranica (Industry)
Responsible Party: Sponsor
Other Study IDs: RWE009
Record Dates: First submitted 2023-11-11; First posted 2023-11-18 (Actual); Results first posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2023-11

CONDITIONS: Migraine
Keywords: REN; Nerivio; Children
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Pre-adolescents with migraine: Patients at the age of 6-11 (included) with migraine who were prescribed the Nerivio device by their healthcare provider and used the Nerivio device at least once
  Interventions: Device: Nerivio

INTERVENTIONS:
Device: Nerivio — Nerivio is a remote electrical neuromodulation (REN) device for the treatment of migraine

SUMMARY:
Migraine is a prevalent neurological disorder that severely impacts both children and adolescents, causing significant disability. Remote Electrical Neuromodulation (REN) is a nonpharmacological, prescribed, wearable device, FDA-cleared for acute and/or preventive treatment of migraine with or without aura in patients 12 years or older. Multiple studies have shown that REN has high safety, tolerability, and efficacy in adults and adolescents. This study aims to evaluate REN's real-world safety and efficacy in pre-adolescents, 6-11 years old.

DETAILED DESCRIPTION:
The REN device (Nerivio by Theranica, Israel) is a neuromodulation device approved by the FDA for acute and/or preventive treatment of migraine in patients 12 years old and above. It is a wearable device applied to the upper arm. It stimulates C and Aδ noxious fibers using a modulated, symmetrical, biphasic, square pulse with a pulse width of 400 μs, modulated frequency of 100-120 Hz, and up to 40 mA output current which the patient can adjust.

The REN device is operated by a designated smartphone application that is downloaded to the user's phone prior first use of the Nerivio device. As part of the sign-up process for the Nerivio app, all patients accept the terms of use which specify that providing personal information is done on their own free will and that their de-identified data may be used for research purposes. Users are not obligated to provide personal information and could treat without providing any feedback. The app includes a secure, personal migraine diary, which enables patients to record and track their migraines attacks and other headaches. At the beginning of each treatment, and again 2 hours after the start of treatment, patients are prompted to record their symptoms, including the presence or absence of aura, pain level (none, mild, moderate, severe), functional disability (none, mild limitation, moderate limitation, severe limitation), presence of associated symptoms (photophobia, phonophobia, and nausea), and an indication of which medications, if any, were taken within that 2-hour time window.

Post-marketing surveillance is designed to assess the safety and efficacy of REN in larger and more diverse populations than in clinical trials and in various real-world environments and situations. As a digital therapeutic device (i.e., electroceutical), the REN device enables prospective collection of electronic patient-reported outcomes in real-world clinical practice.

This post-marketing RWE study investigates the safety and efficacy of the Nerivio treatment in pre-adolescence migraine patients who used the Nerivio device. The following outcomes will be assessed:

1. - Safety - Adverse events that were reported during the study's period
2. - Efficacy - Pain relief, freedom from pain, improvement in functional disability, and improvement in migraine-associated symptoms following the treatment

Together, these objectives provide a comprehensive evaluation of the effect of REN as a treatment for migraine in this target population.

ELIGIBILITY:
Inclusion Criteria:

* Subject age is between 6 to 12 at the date of the REN treatment
* Subject used the Nerivio device at least once

Exclusion Criteria:

* None

Ages: 6 Years to 12 Years | Sex: All
Age Groups: Child
Study Population: Pre-adolescents (age 6-11) who suffer from migraine and use the Nerivio device for acute treatment of migraine.
Sampling Method: Probability Sample
Enrollment: 293 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-05-18 (Actual); Study Completion 2024-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alit Stark-Inbar, PhD, Principal Investigator — Theranica
Locations (2):
- Theranica USA Inc, Bridgewater, New Jersey, United States
- Theranica Bio-Electronics Ltd, Netanya, Israel

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Pre-adolescents With Migraine: Patients at the age of 6-11 (included) with migraines who used the Nerivio device at least once
  Nerivio: Nerivio is a remote electrical neuromodulation (REN) device for the treatment of migraine
Period: Overall Study
Arm/Group | Pre-adolescents With Migraine
Started | 293
Completed | 293
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Pre-adolescents With Migraine
Number analyzed (Participants) | 293
Age, Customized [Count of Participants; unit: Participants] — Age of participants (Years)
  Participants
    11<= and <12 years | 151
    10<= and <11 years | 68
    9<= and <10 years | 34
    8<= and <9 years | 26
    7<= and <8 years | 11
    6<= and <7 years | 3
Sex/Gender, Customized [Count of Participants; unit: Participants] — Baseline measurse were extracted from Nerivio app for each participant Population: Based on the number of participant for each age category
  Participants
    Female (<=11 and <12 years): number analyzed (Participants) | 151
    Female (<=11 and <12 years) | 114
    Female (<=10 Age <11 years): number analyzed (Participants) | 68
    Female (<=10 Age <11 years) | 52
    Female (<=9 and <10 years): number analyzed (Participants) | 34
    Female (<=9 and <10 years) | 21
    Female (<=8 and <9 years): number analyzed (Participants) | 26
    Female (<=8 and <9 years) | 17
    Female (<=7 and <8): number analyzed (Participants) | 11
    Female (<=7 and <8) | 10
    Female (<=6 and <7 years): number analyzed (Participants) | 3
    Female (<=6 and <7 years) | 2
    Male (<=11 and <12 years): number analyzed (Participants) | 151
    Male (<=11 and <12 years) | 37
    Male (<=10 and <11 years): number analyzed (Participants) | 68
    Male (<=10 and <11 years) | 16
    Male (<=9 and <10 years): number analyzed (Participants) | 34
    Male (<=9 and <10 years) | 13
    Male (<=8 and <9 years): number analyzed (Participants) | 26
    Male (<=8 and <9 years) | 9
    Male (<=7 and <8 years): number analyzed (Participants) | 11
    Male (<=7 and <8 years) | 1
    Male (<=6 and <7 years): number analyzed (Participants) | 3
    Male (<=6 and <7 years) | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Rate of Device Related Adverse Events
Description: Incidence of device-related adverse events reported by subjects throughout the study period
Time Frame: Up to 6 months
Measure: Count of Participants; unit: Participants
Groups:
- Pre-adolescence With Migraine: Patients at the age of 6-11 (included) with migraine who used the Nerivio device at least once
  Nerivio: Nerivio is a remote electrical neuromodulation (REN) device for the treatment of migraine
Arm/Group | Pre-adolescence With Migraine
Number analyzed (Participants) | 293
Participants | 0

2. Secondary Outcome: Consistent Headache Relief at 2 Hours Post-treatment
Description: The proportion of subjects reporting headache relief at 2 hours post-treatment in at least 50% of all their treatments.
  Headache relief is defined as an improvement from severe or moderate pain to mild or no pain.
Time Frame: up to 6 months
Population: Patients at the age of 6-11 (included) who used the Nerivio device and had at least 2 pre and post treatments reports were included in the analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-adolescence With Migraine
Number analyzed (Participants) | 18
Participants | 13

3. Secondary Outcome: Consistent Freedom From Headache at 2 Hours Post-treatment
Description: The proportion of subjects reporting freedom from headache at 2 hours post-treatment in at least 50% of all their treatments.
  Pain freedom is defined as the disappearance of headache from severe, moderate, or mild headache at treatment initiation to no headache 2 hours later
Time Frame: up to 6 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-adolescence With Migraine
Number analyzed (Participants) | 25
Participants | 9

4. Secondary Outcome: Consistent Migraine Associated Symptoms Disappearance at 2 Hours Post-treatment
Description: The proportion of subjects reporting the presence of each of the migraine-associated symptoms (nausea/vomiting, photophobia, phonophobia) at the beginning of treatment and reported their absence 2 hours following the treatment in at least 50% of their attacks.
Time Frame: up to 6 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-adolescence With Migraine
Number analyzed (Participants) | 11
Participants
  Nausea/vomiting: number analyzed (Participants) | 10
  Nausea/vomiting | 7
  Photophobia: number analyzed (Participants) | 9
  Photophobia | 2
  Phonophobia: number analyzed (Participants) | 8
  Phonophobia | 4
  At least one symptom | 7

5. Secondary Outcome: Consistent Functional Disability Relief at 2 Hours Post-treatment
Description: The proportion of subjects who reported having Functional Disability at the beginning of the treatment and reported improvement of at least one level of Functional Disability at 2 hours post-treatment in at least 50% of all their treatments.
Time Frame: up to 6 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Groups:
- Pre-adolescence With Migraine: Patients at the age of 6-11 (included) with migraines who used the Nerivio device at least once
  Nerivio: Neriio is a remote electrical neuromodulation (REN) device for the treatment of migraine
Arm/Group | Pre-adolescence With Migraine
Number analyzed (Participants) | 18
Participants | 15

6. Secondary Outcome: Consistent Functional Disability Disappearance at 2 Hours Post-treatment
Description: The proportion of subjects who reported having Functional Disability at the beginning of the treatment and reported no Functional Disability at 2 hours post-treatment in at least 50% of all their treatments.
Time Frame: up to 6 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-adolescence With Migraine
Number analyzed (Participants) | 18
Participants | 7

ADVERSE EVENTS:
Time Frame: Up to 7 months
Groups:
- Pre-adolescence With Migraine: Patients at the age of 6-12 with migraines who used the Nerivio device at least once
  Nerivio: Neriio is a remote electrical neuromodulation (REN) device for the treatment of migraine
Arm/Group | Pre-adolescence With Migraine
All-Cause Mortality (participants affected / at risk) | 0/293
Serious Adverse Events (participants affected / at risk) | 0/293
Other Adverse Events (participants affected / at risk) | 0/293

LIMITATIONS AND CAVEATS:
A post-marketing cohort study without a control group; not all participants provided data for efficacy calculations; age among the cohort of children is not uniformly distributed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-02-10): https://cdn.clinicaltrials.gov/large-docs/56/NCT06138756/Prot_SAP_000.pdf